CLINICAL TRIAL: NCT07153406
Title: Comparison of Esketamine Versus Aripiprazole,Both in Combination With a SSRI/SNRI(Selective Serotonin Reuptake Inhibitors/Serotonin and Norepinephrine Reuptake Inhibitors )in Treatment-resistant Major Depressive Disorder in Elderly Patients
Brief Title: Comparison of Esketamine Nasal Spray vs.Aripiprazole in Treat.Resistant Major Depressive Disorder in Elderly Patients
Acronym: CESAR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CESAR
Record Dates: First submitted 2024-10-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder
Keywords: Depressive Disorder; Moderate-severe depressive episode.; Antidepressants; Psychotropics
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blind for evaluators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine (Experimental): Esketamine intranasal spray at flexible doses 28, 56 and 84 mg once or twice a week
  Interventions: Drug: Experimental regimen
- aripiprazole (Active Comparator): Oral aripiprazole 5-30 mg daily, once or twice daily for the duration of the study
  Interventions: Drug: Control regimen

INTERVENTIONS:
Drug: Experimental regimen — Esketamine intranasal spray at flexible doses (28, 56 and 84 mg) once or twice a week
  Arms: Esketamine
Drug: Control regimen — Oral aripiprazole 5-30 mg daily, once or twice daily for the duration of the study
  Arms: aripiprazole

SUMMARY:
Phase III, open label, randomised, multicentre, blind for evaluators clinical trial to evaluate the efficacy of esketamine nasal spray at flexible dosis compared to aripiprazole in elderly participants (>60 years) who suffer from treatment-resistant major depressive

DETAILED DESCRIPTION:
The study disease is resistant major depressive disorder, which has not responded to at least three different strategies with antidepressants, at least one of them being a combination or potentiation strategy, with a current moderate-severe depressive episode.

The aim of the study is to evaluate the efficacy of esketamine nasal spray at flexible dosis compared to aripiprazole at 8 weeks, both in combination with a continued antidepressant, in elderly participants (>60 years), who suffer from treatment-resistant major depressive disorder with one episode current moderate to severe depressive disorder

ELIGIBILITY:
Inclusion Criteria:

* Patients between 60-74 years
* To be receiving antidepressant treatment that includes an antidepressant at the time of screening that is not responding (less than 25% improvement in symptoms) after receiving an adequate dose [or local equivalent, if applicable] for at least 6 weeks and have been increased to the dose maximum allowed
* Current antidepressant treatment must have been immediately preceded by failure to respond to at least 3, but not more than 5, different consecutive treatments (all within the same moderately severe depressive episode) with antidepressant drugs (AD) taken at an appropriate dose for at least least 6 weeks (3 antidepressant failures including the current one)
* To have been treated with at least 3 different classes of antidepressants between treatments taken at appropriate doses for at least 6 weeks without response in the current moderate to severe depressive episode (including current treatment with an antidepressant)
* To be taking a single oral antidepressant on day 1 before randomization
* Participants who, at the time of screening, are taking a combination of antidepressants and/or rescue treatment (other than aripiprazole) for the current moderate to severe depressive episode may participate in the study.

Exclusion Criteria:

* Treatment with drugs contraindicated with the use of esketamine and aripiprazole.
* Patients in whom a high risk of suicide is detected at the screening visit, according to the criteria established by Columbia University according to the C-SSRS evaluation
* Patients who are participating in another clinical trial with active treatment
* Patients who do not have the capacity to consent to participation in the trial or who do not have a representative to confirm their participation
* Hypersensitivity to any of the active ingredients of any of the branches of treatment, or to any of the excipients of its pharmaceutical form
* Patients in whom increased blood pressure or blood pressure intracranial fluid poses a serious risk

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Clinical response | At week 8
  Clinical response at week 8 after initiation of treatment, measured in terms of:
  * Remission of depressive symptoms; total score ≤10 on the MADRS (Montgomery-Asberg Depression Rating Scale )scale.
  * Adequate clinical response, if they show a reduction of ≥50% in the total score of the MADRS scale with respect to the initial score and a score ≤4 on the CGI severity scale. (Clinical Global Impression)

SECONDARY OUTCOMES:
Safety profile of esketamine nasal spray and aripiprazole | At week 32
  Determination of the safety profile of esketamine nasal spray and aripiprazole in patients free of relapse at week 32, according to the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 throughout the study.
Clinical response | At week 32
  Clinical response measured in terms of:
  * Remission of depressive symptoms; total score ≤10 on the MADRS scale.
  * Adequate clinical response, if they show a reduction of ≥50% in the total score of the MADRS scale compared to the initial score and a score ≤4 on the CGI severity scale.
Safety profile of esketamine nasal spray and aripiprazole | At week 8
  Determination of the safety profile of esketamine nasal spray and aripiprazole at week 8, according to the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 throughout the study.
Free of relapse | At week 24, at week 32
  Proportion of patients free of relapse at week 24 and week 32 in the group of patients with clinical remission at week 8.
Score on the EuroQol-5D scale (www.euroqol.org) | At day 1, at day 8, at day 15, at day 22, at week 5 to 8, at week 9 to 32, at week 34
  Score on the EuroQol-5D (EQ-5D) health-related quality of life scale in adults
Obtaining the transcriptome | At week 8, at week 32
  Obtaining the transcriptome of patients at week 8 and week 32 of treatment using a large-scale sequencer.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo Facorro, MD, Principal Investigator — Fundación para la Gestión de la Investigación en Salud de Sevilla
Locations (9):
- Spain (9):
  - Clínica Psiquiátrica Padre Menni, Pamplona, Navarre
  - Hospital Vall d'Hebron, Barcelona
  - Hospital De La Santa Creu i Sant Pau, Barcelona
  - Hospital Mare de Déu de La Mercè, Barcelona
  - Hospital Sagrat Cor. Martorell, Barcelona
  - Hospital Benito Menni y Fidmag Hermanas Hospitalarias, Barcelona
  - Centro Sociosanitario Hermanas Hospitalarias de Palencia, Palencia
  - Corporacion Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville